CLINICAL TRIAL: NCT04482075
Title: Cross-modality Matching Between Pressure Pain Threshold and Subjective Ratings of Pain Intensity, Affect and Disability in Patients With Chronic Low Back Pain.
Brief Title: Relationship Between Pressure Pain Threshold and Pain Intensity, Affect and Disability in CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00002
Record Dates: First submitted 2020-02-22; First posted 2020-07-22 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Pain Threshold; Low Back Pain; Pain Measurement
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SEGMENTAL STABILISATION TRAINING (SST) (Other): Segmental Stabilisation Training is an established treatment technique for chronic low back pain
  Interventions: Other: segmental stability training

INTERVENTIONS:
Other: segmental stability training — SEGMENTAL STABILISATION TRAINING (SST): This part of the therapy shall involve Isometric co-contraction of Lumbar Transversus abdominis and Lumbar Multifidus. The patient shall perform 10 repetitions of abdominal drawing-in manoeuvre with 30-40% Maximal Voluntary Contraction (MVC) with a 10-second hold in specific prescribed positions.

SUMMARY:
The association between pressure pain threshold and different aspects of low back pain has garnered attention over the years. However, since most of such studies in the past employed cross sectional designs, a longitudinal study design with follow-up measurements is required to further investigate this relationship. Studying this relationship will not only offer insights into the phenomenon of pain but may also bring us one step closer to achieving the seemingly insurmountable goal of objectively measuring back pain and its different dimensions.

DETAILED DESCRIPTION:
This study is aimed to examine and evaluate the true extent of the relationship between pressure pain threshold (PPT) and different aspects of somatic pain, by studying the interplay between PPT and different variables, and by further exploring the predictive capability of PPT values to estimate pain intensity, pain affect and disability associated with chronic low back pain (CLBP). In order to estimate these dimensions a calculator based on mathematical equations using different predictive models will be developed. This tool (calculator) will take into account PPT reading from the lower back region and some other variables having confounding effects on PPT and pain, and will be able to predict pain intensity, affect and associated disability with reasonable accuracy. Patients with chronic low back pain shall be the target population and shall be recruited through referrals from the medical Out-Patients Department of Institute of Physical Medicine & Rehabilitation, Dow University of Health Sciences and Department of Rehabilitation Medicine PNS-Shifa Hospital, Karachi, Pakistan after initial screening in accordance with the inclusion and exclusion criteria. Screened patients shall then be briefed about the research project. After explaining the study objectives, procedures, potential benefits and discomforts, written informed consent shall be obtained from the patients. Only upon their agreement shall they become study participants and undergo assessments. The study participants shall receive handouts to document Depression and Anxiety, Pain Intensity, Pain Affect, and Disability. Pressure pain threshold (PPT) shall be measured using a manual Algometer. These measurements shall be followed by a session of physiotherapy treatment, after which Pain Intensity, Pain Affect, and Disability shall be recorded again.

ELIGIBILITY:
Inclusion Criteria:

* Adult males with low back pain with an age group of 18-50 years.

Exclusion Criteria:

1. Individuals having low back pain for less than 3 months.
2. Individuals with specific underlying pathology as the cause of CLBP. (Active oncological disease, Known disc derangement, cauda equina syndrome, spinal trauma i.e. fracture, neuropathy i.e. sciatica or severe root compression, spinal structural deformity, infection, inﬂammatory joint disease, spinal stenosis, spondylolysis, spondylolisthesis).
3. Individuals having neurological diseases (including central and peripheral diseases); metabolic diseases (i.e. diabetes and hypothyroidism); coagulopathies (i.e. haemophilia).
4. Individuals with fibromyalgia syndrome (FMS); myofascial pain syndrome (MPS); allodynia (stroking hyperalgesia).
5. Individuals suffering from aphasia or suffering from deafness, blindness or muteness.
6. Individuals with skin disease (i.e. psoriasis, scleroderma, leprosy, etc.) or skin lesions (i.e. abrasion/laceration/ bruise) in the low back region.
7. Individuals having oral temperature of 100 F or above.
8. Individuals who have undergone spinal surgery.
9. Individuals scoring 28+ for depression, 20+ for anxiety, 34+ for stress on DASS-21.
10. Individuals in whom prone lying causes significant discomfort (i.e. dyspnoea etc.).
11. Individuals who do not perceive pressure pain below 10 kg/cm2 during PPT testing.
12. Individuals evincing bruising to PPT testing.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult males with low back pain with an age group of 18-50 years.
Enrollment: 41 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Pressure threshold meter | Up to 2 weeks
  Its a type of force gauge which consists of a rubber-tipped plunger with a surface area of usually 1cm square, connected to the force gauge (body) via a metal rod. The force gauge is usually calibrated in Newtons or Kilograms per cm2 with a range of up to 10 kgs. The exerted pressure on the plunger is transmitted to the gauge through the metal rod, which in turn moves the indicator needle in the clockwise direction with a magnitude corresponding to the force applied. The indicator needle remains in this position until the zeroing knob is pressed, which brings the needle back to its starting position. This allows the examiner to record the last reading of the pressure applied after removing the device from the body.
Visual Analogue scale (VAS) - pain intensity | Up to 2 weeks
  Visual Analogue scale furnished with specific anchors to measure pain intensity. It is a continuous scale that is considered as a unidimensional measure of the pain experience. It consists of a 100 mm straight line, anchored by descriptors such as 'no pain at all' (0mm) and 'worst pain imaginable' (100mm) at both extremes. The respondent marks the line which corresponds to the current state of pain. Scoring is done with the help of a ruler and the whole process takes about a minute to complete. VAS demonstrates ratio-scale properties and it can be adapted to assess dimensions other than intensity such as unpleasantness (affective dimension) associated with pain.
Visual Analogue scale (VAS) - pain affect | Up to 2 weeks
  Visual analogue scale fine-tuned to measure pain affect with specific anchors. In general, the same technique used for assessing the pain intensity may be used to assess the pain affect. It consists of a 100 mm straight line, anchored by descriptors such as ''not bad at all'' (0mm) and ''the most unpleasant feeling possible for me'' (100mm) at both extremes. The respondent marks the line which corresponds to the current state of pain. Scoring is done with the help of a ruler and the whole process takes about a minute to complete.
Disability Rating Index (DRI) | Up to 2 weeks
  This article focuses on the Disability Rating Index (DRI), a patient-reported outcome measure developed by Salén et al. in 1994, with the aim of measuring the physical disability of respondents within a clinical setting. The DRI evaluates a respondent's disability by assessing activity and participation limitations. It covers 12 non-specific activities of daily life, each one self-rated on a visual analogue scale of 0-100 mm, providing a score of 0-100 for each activity, where 0 represents no difficulty in performing the specific task and 100 indicates an inability to perform the task at all.

SECONDARY OUTCOMES:
Saltin-Grimby Physical Activity Level Scale (SGPALS) | At baseline
  It's a four-level questionnaire to assess leisure-time physical activity (PA). It is anchored by descriptors such as "physically inactive" (0) and "regular hard physical training for competitive sports" (4).
Depression, Anxiety and Stress Scale (DASS-21) | Up to 2 weeks
  This is a set of three self-report scales designed to measure the emotional states of depression, anxiety & stress. The minimum score lies between 0 - 3 (normal) and the maximum score 14 and above (Extremely Severe). For Anxiety 0 - 3 (normal) and the maximum score 10 and above (Extremely Severe) and For Stress 0 - 7 (normal) and the maximum score 17 and above (Extremely Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Rasim Ul Hasanat Qureshi, MSPT, Principal Investigator — Dow University of Health Sciences; Shahzad Ali Syed, MSAPT, Study Director — Dow University of Health Sciences
Locations (1):
- Institute of Physical medicine & Rehabilitation, Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Ul Hasanat R, Syed SA, Rathore FA, Iftikhar S. Development of a tool for objectively measuring somatic pain in the low back region based on a longitudinal diagnostic study conducted in Karachi, Pakistan. BMJ Open. 2023 Mar 16;13(3):e067129. doi: 10.1136/bmjopen-2022-067129. PMID 36927595